CLINICAL TRIAL: NCT02134028
Title: Open-label Extension Study to Evaluate the Long-term Safety and Tolerability of Dupilumab in Patients With Asthma Who Participated in a Previous Dupilumab Asthma Clinical Study
Brief Title: Long-Term Safety Evaluation of Dupilumab in Patients With Asthma (LIBERTY ASTHMA TRAVERSE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS12551; 2013-003856-19 (EudraCT Number); U1111-1117-6745 (Other: UTN)
Record Dates: First submitted 2014-04-30; First posted 2014-05-08 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- dupilumab treatment (Experimental): For participants coming from the DRI12544 study: dupilumab loading dose subcutaneous (SC) on Day 1, followed by 1* Dose every 2 weeks added to current controller medications.
  For participants coming from other studies: dupilumab 1 * Dose SC every 2 weeks added to current controller medications.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Pharmaceutical form: Solution for injection Routes of administration: Subcutaneous
  Other Names: SAR231893; REGN668

SUMMARY:
Primary Objective:

To evaluate the long-term safety and tolerability of dupilumab in participants with asthma who participated in a previous dupilumab asthma study (DRI12544, PDY14192, EFC13579, EFC13691).

Secondary Objectives:

To evaluate the long-term efficacy of dupilumab in participants with asthma who participated in a previous dupilumab asthma clinical study.

To evaluate dupilumab in participants with asthma who participated in a previous dupilumab asthma clinical study, with regards to:

* Systemic exposure
* Anti-drug antibodies
* Biomarkers

DETAILED DESCRIPTION:
A screening period, up to 3 weeks, applied only for participants who came from DRI12544 study. The total study duration, per participant, was a maximum of 108 weeks (or 111 weeks considering a maximum screening period of 3 weeks for study DRI12544) for the participants enrolled prior to Amendment 04 approval and a maximum of 60 weeks for the participants enrolled after Amendment 04 approval.

Following amendment 04 (dated 31 Oct 2016) the open-label treatment duration was amended to 48 weeks (1 year); and the 16-week post-treatment period was shortened to 12 weeks.

ELIGIBILITY:
Inclusion criteria:

- Participants with asthma who completed the treatment period in a previous dupilumab asthma clinical study (i.e., PDY14192, EFC13579 or EFC13691) or participants with asthma who completed the treatment and follow-up periods in previous dupilumab asthma Study DRI12544.

Exclusion criteria:

- Participants who experienced any hypersensitivity reactions to Investigational Medicinal Product (IMP) in the previous dupilumab asthma study, which, in the opinion of the Investigator, could indicate that continued treatment with dupilumab, may present an unreasonable risk for the participant.

The above information was not intended to contain all considerations relevant to a Participant's potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2282 (Actual)
Dates: Start 2014-08-05 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (365):
- United States (82):
  - Investigational Site Number 840047, Birmingham, Alabama
  - Investigational Site Number 840099, Gilbert, Arizona
  - Investigational Site Number 840087, Scottsdale, Arizona
  - Investigational Site Number 840402, Tucson, Arizona
  - Investigational Site Number 840132, Little Rock, Arkansas
  - Investigational Site Number 840109, Bakersfield, California
  - Investigational Site Number 840045, Long Beach, California
  - Investigational Site Number 840019, Los Angeles, California
  - Investigational Site Number 840029, Los Angeles, California
  - Investigational Site Number 840022, Los Angeles, California
  - Investigational Site Number 840044, Newport Beach, California
  - Investigational Site Number 840041, North Hollywood, California
  - Investigational Site Number 840014, Rolling Hills Estates, California
  - Investigational Site Number 840121, San Jose, California
  - Investigational Site Number 840040, Colorado Springs, Colorado
  - Investigational Site Number 840403, Denver, Colorado
  - Investigational Site Number 840006, Denver, Colorado
  - Investigational Site Number 840024, Denver, Colorado
  - Investigational Site Number 840130, Denver, Colorado
  - Investigational Site Number 840902, New Haven, Connecticut
  - Investigational Site Number 840137, Aventura, Florida
  - Investigational Site Number 840071, Gainesville, Florida
  - Investigational Site Number 840115, Ocoee, Florida
  - Investigational Site Number 840055, Sarasota, Florida
  - Investigational Site Number 840079, Twin Falls, Idaho
  - Investigational Site Number 840101, Chicago, Illinois
  - Investigational Site Number 840032, Fort Mitchell, Kentucky
  - Investigational Site Number 840017, Louisville, Kentucky
  - Investigational Site Number 840030, Owensboro, Kentucky
  - Investigational Site Number 840064, Bangor, Maine
  - Investigational Site Number 840052, Chevy Chase, Maryland
  - Investigational Site Number 840073, Gaithersburg, Maryland
  - Investigational Site Number 840080, Owings Mills, Maryland
  - Investigational Site Number 840401, Boston, Massachusetts
  - Investigational Site Number 840018, Minneapolis, Minnesota
  - Investigational Site Number 840002, St Louis, Missouri
  - Investigational Site Number 840102, St Louis, Missouri
  - Investigational Site Number 840093, St Louis, Missouri
  - Investigational Site Number 840037, Missoula, Montana
  - Investigational Site Number 840078, Omaha, Nebraska
  - Investigational Site Number 840004, Papillion, Nebraska
  - Investigational Site Number 840111, Brick, New Jersey
  - Investigational Site Number 840068, Ocean City, New Jersey
  - Investigational Site Number 840011, Princeton, New Jersey
  - Investigational Site Number 840065, New York, New York
  - Investigational Site Number 840126, Charlotte, North Carolina
  - Investigational Site Number 840083, Charlotte, North Carolina
  - Investigational Site Number 840108, Durham, North Carolina
  - Investigational Site Number 840107, Greensboro, North Carolina
  - Investigational Site Number 840907, High Point, North Carolina
  - Investigational Site Number 840404, Winston-Salem, North Carolina
  - Investigational Site Number 840015, Cincinnati, Ohio
  - Investigational Site Number 840146, Cincinnati, Ohio
  - Investigational Site Number 840049, Middleburg Heights, Ohio
  - Investigational Site Number 840942, Toledo, Ohio
  - Investigational Site Number 840112, Edmond, Oklahoma
  - Investigational Site Number 840104, Tulsa, Oklahoma
  - Investigational Site Number 840034, Medford, Oregon
  - Investigational Site Number 840031, Portland, Oregon
  - Investigational Site Number 840046, Bethlehem, Pennsylvania
  - Investigational Site Number 840085, Hershey, Pennsylvania
  - Investigational Site Number 840067, Philadelphia, Pennsylvania
  - Investigational Site Number 840928, Pittsburgh, Pennsylvania
  - Investigational Site Number 840091, Pittsburgh, Pennsylvania
  - Investigational Site Number 840082, Charleston, South Carolina
  - Investigational Site Number 840117, Greenville, South Carolina
  - Investigational Site Number 840021, Spartanburg, South Carolina
  - Investigational Site Number 840062, Amarillo, Texas
  - Investigational Site Number 840038, Boerne, Texas
  - Investigational Site Number 840124, Cypress, Texas
  - Investigational Site Number 840023, Dallas, Texas
  - Investigational Site Number 840923, El Paso, Texas
  - Investigational Site Number 840922, Fort Worth, Texas
  - Investigational Site Number 840027, Fort Worth, Texas
  - Investigational Site Number 840070, McKinney, Texas
  - Investigational Site Number 840118, Plano, Texas
  - Investigational Site Number 840008, San Antonio, Texas
  - Investigational Site Number 840035, Draper, Utah
  - Investigational Site Number 840077, Murray, Utah
  - Investigational Site Number 840057, South Burlington, Vermont
  - Investigational Site Number 840059, Fairfax, Virginia
  - Investigational Site Number 840951, Bellingham, Washington
- Argentina (15):
  - Investigational Site Number 032096, Bahía Blanca
  - Investigational Site Number 032004, Buenos Aires
  - Investigational Site Number 032003, Buenos Aires
  - Investigational Site Number 032011, Caba
  - Investigational Site Number 032097, Caba
  - Investigational Site Number 032001, Caba
  - Investigational Site Number 032010, Caba
  - Investigational Site Number 032091, Caba
  - Investigational Site Number 032095, Capital Federal
  - Investigational Site Number 032002, La Plata
  - Investigational Site Number 032006, Rosario
  - Investigational Site Number 032007, Rosario
  - Investigational Site Number 032005, Rosario
  - Investigational Site Number 032012, San Miguel de Tucumán
  - Investigational Site Number 032009, San Miguel de Tucumán
- Australia (9):
  - Investigational Site Number 036004, Adelaide
  - Investigational Site Number 036005, Campbelltown
  - Investigational Site Number 036001, Clayton
  - Investigational Site Number 036008, Frankston
  - Investigational Site Number 036093, Murdoch
  - Investigational Site Number 036003, Nedlands
  - Investigational Site Number 036094, Parkville
  - Investigational Site Number 036009, Prahran
  - Investigational Site Number 036006, Woolloongabba
- Belgium (3):
  - Investigational Site Number 056002, Brussels
  - Investigational Site Number 056003, Ghent
  - Investigational Site Number 056001, Leuven
- Brazil (8):
  - Investigational Site Number 076009, Florianópolis
  - Investigational Site Number 076007, Porto Alegre
  - Investigational Site Number 076001, Porto Alegre
  - Investigational Site Number 076003, Salvador
  - Investigational Site Number 076013, São Bernardo do Campo
  - Investigational Site Number 076012, São Paulo
  - Investigational Site Number 076006, São Paulo
  - Investigational Site Number 076002, Sorocaba
- Canada (16):
  - Investigational Site Number 124019, Burlington
  - Investigational Site Number 124009, Calgary
  - Investigational Site Number 124016, Hamilton
  - Investigational Site Number 124003, Mississauga
  - Investigational Site Number 124001, Montreal
  - Investigational Site Number 124012, Montreal
  - Investigational Site Number 124010, Montreal
  - Investigational Site Number 124013, Ottawa
  - Investigational Site Number 124018, Québec
  - Investigational Site Number 124014, Québec
  - Investigational Site Number 124008, Sherbrooke
  - Investigational Site Number 124015, Toronto
  - Investigational Site Number 124002, Toronto
  - Investigational Site Number 124007, Trois-Rivières
  - Investigational Site Number 124006, Vancouver
  - Investigational Site Number 124017, Vancouver
- Chile (14):
  - Investigational Site Number 152007, Quillota
  - Investigational Site Number 152024, Santiago
  - Investigational Site Number 152005, Santiago
  - Investigational Site Number 152014, Santiago
  - Investigational Site Number 152011, Santiago
  - Investigational Site Number 152018, Santiago
  - Investigational Site Number 152002, Santiago
  - Investigational Site Number 152013, Santiago
  - Investigational Site Number 152008, Talca
  - Investigational Site Number 152004, Talca
  - Investigational Site Number 152023, Talcahuano
  - Investigational Site Number 152010, Valdivia
  - Investigational Site Number 152003, Viña del Mar
  - Investigational Site Number 152021, Viña del Mar
- Colombia (2):
  - Investigational Site Number 170001, Bogotá
  - Investigational Site Number 170002, Bogotá
- Denmark (2):
  - Investigational Site Number 208002, Hvidovre
  - Investigational Site Number 208001, København NV
- France (11):
  - Investigational Site Number 250009, Brest
  - Investigational Site Number 250004, La Tronche
  - Investigational Site Number 250010, Lille
  - Investigational Site Number 250013, Lille
  - Investigational Site Number 250006, Lyon
  - Investigational Site Number 250001, Marseille
  - Investigational Site Number 250002, Montpellier
  - Investigational Site Number 250005, Nantes
  - Investigational Site Number 250007, Nîmes
  - Investigational Site Number 250008, Strasbourg
  - Investigational Site Number 250014, Vandœuvre-lès-Nancy
- Germany (6):
  - Investigational Site Number 276006, Berlin
  - Investigational Site Number 276003, Bochum
  - Investigational Site Number 276010, Frankfurt am Main
  - Investigational Site Number 276011, Großhansdorf
  - Investigational Site Number 276009, Koblenz
  - Investigational Site Number 276005, Rüdersdorf Bei Berlin
- Hungary (3):
  - Investigational Site Number 348301, Balassagyarmat
  - Investigational Site Number 348303, Edelény
  - Investigational Site Number 348003, Gödöllö
- Israel (4):
  - Investigational Site Number 376003, Haifa
  - Investigational Site Number 376001, Kfar Saba
  - Investigational Site Number 376005, Petah Tikva
  - Investigational Site Number 376002, Rehovot
- Italy (9):
  - Investigational Site Number 380010, Ancona
  - Investigational Site Number 380009, Catania
  - Investigational Site Number 380004, Ferrara
  - Investigational Site Number 380008, Foggia
  - Investigational Site Number 380002, Genova
  - Investigational Site Number 380003, Modena
  - Investigational Site Number 380007, Padua
  - Investigational Site Number 380099, Palermo
  - Investigational Site Number 380001, Pisa
- Japan (62):
  - Investigational Site Number 392185, Akashi-Shi
  - Investigational Site Number 392009, Asahi-Shi
  - Investigational Site Number 392037, Chiyoda-Ku
  - Investigational Site Number 392002, Chūōku
  - Investigational Site Number 392007, Chūōku
  - Investigational Site Number 392112, Chūōku
  - Investigational Site Number 392012, Edogawa-Ku
  - Investigational Site Number 392137, Fukuoka
  - Investigational Site Number 392021, Fukuyama-Shi
  - Investigational Site Number 392030, Habikino-Shi
  - Investigational Site Number 392004, Himeji-Shi
  - Investigational Site Number 392032, Hirakata-Shi
  - Investigational Site Number 392108, Hiroshima
  - Investigational Site Number 392158, Hiroshima
  - Investigational Site Number 392013, Iizuka-Shi
  - Investigational Site Number 392042, Isesaki-Shi
  - Investigational Site Number 392023, Kanazawa
  - Investigational Site Number 392142, Kasuga-Shi
  - Investigational Site Number 392119, Kishiwada-Shi
  - Investigational Site Number 392025, Kobe
  - Investigational Site Number 392162, Kobe
  - Investigational Site Number 392040, Kodaira-Shi
  - Investigational Site Number 392044, Kokubunji-Shi
  - Investigational Site Number 392131, Koushi-Shi
  - Investigational Site Number 392010, Kurashiki-Shi
  - Investigational Site Number 392036, Kyoto
  - Investigational Site Number 392153, Kyoto
  - Investigational Site Number 392133, Machida-Shi
  - Investigational Site Number 392135, Matsuyama
  - Investigational Site Number 392122, Minatoku
  - Investigational Site Number 392144, Minatoku
  - Investigational Site Number 392106, Mizunami-Shi
  - Investigational Site Number 392164, Muroran-Shi
  - Investigational Site Number 392163, Nagoya
  - Investigational Site Number 392020, Naka-Gun
  - Investigational Site Number 392005, Naruto-Shi
  - Investigational Site Number 392187, Obihiro-Shi
  - Investigational Site Number 392177, Ome-Shi
  - Investigational Site Number 392152, Osaka Sayama-Shi
  - Investigational Site Number 392155, Osaka Sayama-Shi
  - Investigational Site Number 392170, Osaki-Shi
  - Investigational Site Number 392043, Ota-Shi
  - Investigational Site Number 392127, Ōta-ku
  - Investigational Site Number 392169, Sagamihara-Shi
  - Investigational Site Number 392011, Sakaide-Shi
  - Investigational Site Number 392024, Sakaishi
  - Investigational Site Number 392008, Sapporo
  - Investigational Site Number 392034, Sapporo
  - Investigational Site Number 392038, Setagaya-Ku
  - Investigational Site Number 392179, Seto-Shi
  - Investigational Site Number 392186, Shibuya-Ku
  - Investigational Site Number 392167, Shinagawa-Ku
  - Investigational Site Number 392130, Shinjuku-Ku
  - Investigational Site Number 392165, Sumida-Ku
  - Investigational Site Number 392146, Tachikawa-Shi
  - Investigational Site Number 392173, Tachikawa-Shi
  - Investigational Site Number 392006, Tomakomai-Shi
  - Investigational Site Number 392029, Tsu
  - Investigational Site Number 392168, Uozu-Shi
  - Investigational Site Number 392132, Urasoe-Shi
  - Investigational Site Number 392045, Uruma
  - Investigational Site Number 392014, Yokohama
- Mexico (12):
  - Investigational Site Number 484013, Chihuahua City
  - Investigational Site Number 484006, Chihuahua City
  - Investigational Site Number 484014, Cuautitlán Izcalli
  - Investigational Site Number 484005, Distrito Federal
  - Investigational Site Number 484008, Durango
  - Investigational Site Number 484001, Guadalajara
  - Investigational Site Number 484004, Mexico City
  - Investigational Site Number 484010, México
  - Investigational Site Number 484003, Monterrey
  - Investigational Site Number 484007, Monterrey
  - Investigational Site Number 484012, San Juan del Río
  - Investigational Site Number 484011, Veracruz
- Netherlands (2):
  - Investigational Site Number 528001, Arnhem
  - Investigational Site Number 528002, Dordrecht
- Poland (13):
  - Investigational Site Number 616006, Bialystok
  - Investigational Site Number 616004, Gdansk
  - Investigational Site Number 616003, Gdansk
  - Investigational Site Number 616007, Krakow
  - Investigational Site Number 616097, Krakow
  - Investigational Site Number 616001, Lodz
  - Investigational Site Number 616005, Lodz
  - Investigational Site Number 616009, Lodz
  - Investigational Site Number 616096, Poznan
  - Investigational Site Number 616098, Strzelce Opolskie
  - Investigational Site Number 616008, Warsaw
  - Investigational Site Number 616010, Warsaw
  - Investigational Site Number 616011, Żnin
- Romania (6):
  - Investigational Site Number 642104, Bucharest
  - Investigational Site Number 642103, Bucharest
  - Investigational Site Number 642102, Cluj-Napoca
  - Investigational Site Number 642107, Cluj-Napoca
  - Investigational Site Number 642105, Timișoara
  - Investigational Site Number 642106, Timișoara
- Russia (14):
  - Investigational Site Number 643096, Moscow
  - Investigational Site Number 643002, Moscow
  - Investigational Site Number 643005, Moscow
  - Investigational Site Number 643007, Moscow
  - Investigational Site Number 643012, Moscow
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643006, Novosibirsk
  - Investigational Site Number 643091, Ryazan
  - Investigational Site Number 643099, Saint Petersburg
  - Investigational Site Number 643011, Saint Petersburg
  - Investigational Site Number 643010, Saint Petersburg
  - Investigational Site Number 643009, Saint Petersburg
  - Investigational Site Number 643008, Yaroslavl
  - Investigational Site Number 643013, Yekaterinburg
- South Africa (9):
  - Investigational Site Number 710011, Cape Town
  - Investigational Site Number 710001, Cape Town
  - Investigational Site Number 710091, Cape Town
  - Investigational Site Number 710092, Cape Town
  - Investigational Site Number 710002, Cape Town
  - Investigational Site Number 710003, Cape Town
  - Investigational Site Number 710006, Durban
  - Investigational Site Number 710007, Pretoria
  - Investigational Site Number 710009, Winnie Mandela
- South Korea (12):
  - Investigational Site Number 410002, Bucheon-si
  - Investigational Site Number 410003, Cheongju-si
  - Investigational Site Number 410013, Incheon
  - Investigational Site Number 410006, Seoul
  - Investigational Site Number 410008, Seoul
  - Investigational Site Number 410004, Seoul
  - Investigational Site Number 410012, Seoul
  - Investigational Site Number 410005, Seoul
  - Investigational Site Number 410007, Seoul
  - Investigational Site Number 410010, Seoul
  - Investigational Site Number 410011, Seoul
  - Investigational Site Number 410001, Suwon
- Spain (10):
  - Investigational Site Number 724014, Barcelona
  - Investigational Site Number 724002, Barcelona
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724010, Palma de Mallorca
  - Investigational Site Number 724006, Pozuelo de Alarcón
  - Investigational Site Number 724003, Sabadell
  - Investigational Site Number 724007, Sant Boi de Llobregat
  - Investigational Site Number 724096, Santiago de Compostela
  - Investigational Site Number 724008, Seville
  - Investigational Site Number 724097, Valencia
- Taiwan (3):
  - Investigational Site Number 158008, New Taipei City
  - Investigational Site Number 158007, Taichung
  - Investigational Site Number 158009, Taipei
- Turkey (Türkiye) (12):
  - Investigational Site Number 792002, Ankara
  - Investigational Site Number 792098, Ankara
  - Investigational Site Number 792008, Bursa
  - Investigational Site Number 792007, Istanbul
  - Investigational Site Number 792001, Istanbul
  - Investigational Site Number 792004, Istanbul
  - Investigational Site Number 792003, Istanbul
  - Investigational Site Number 792005, Izmir
  - Investigational Site Number 792090, Izmir
  - Investigational Site Number 792013, Kırıkkale
  - Investigational Site Number 792006, Mersin
  - Investigational Site Number 792096, Rize
- Ukraine (21):
  - Investigational Site Number 804007, Chernivtsi
  - Investigational Site Number 804023, Dnipro
  - Investigational Site Number 804009, Ivano-Frankivsk
  - Investigational Site Number 804094, Ivano-Frankivsk
  - Investigational Site Number 804005, Kharkiv
  - Investigational Site Number 804021, Kharkiv
  - Investigational Site Number 804001, Kharkiv
  - Investigational Site Number 804004, Kyiv
  - Investigational Site Number 804003, Kyiv
  - Investigational Site Number 804008, Kyiv
  - Investigational Site Number 804017, Kyiv
  - Investigational Site Number 804018, Kyiv
  - Investigational Site Number 804020, Kyiv
  - Investigational Site Number 804016, Kyiv
  - Investigational Site Number 804006, Odesa
  - Investigational Site Number 804002, Poltava
  - Investigational Site Number 804014, Ternopil
  - Investigational Site Number 804019, Vinnytsia
  - Investigational Site Number 804015, Yalta
  - Investigational Site Number 804022, Zaporizhzhya
  - Investigational Site Number 804012, Zaporizhzhya
- United Kingdom (5):
  - Investigational Site Number 826001, Bradford
  - Investigational Site Number 826010, London
  - Investigational Site Number 826009, Oxford
  - Investigational Site Number 826007, Portsmouth
  - Investigational Site Number 826006, South Shields

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Pavord ID, Wechsler ME, Busse WW, Domingo C, Xia C, Gall R, Pandit-Abid N, Jacob-Nara JA, Radwan A, Rowe PJ, Deniz Y. Dupilumab efficacy in patients with type 2 asthma and early Feno level reductions. J Allergy Clin Immunol Glob. 2025 Apr 15;4(3):100474. doi: 10.1016/j.jacig.2025.100474. eCollection 2025 Aug. PMID 40458676
- [Derived] Rhee CK, Park JW, Park HW, Noh H, Msihid J, Cho YS. Long-term Safety and Efficacy of Dupilumab in Patients With Uncontrolled, Moderate-to-Severe Asthma Recruited From Korean Centers: A Subgroup Analysis of the Phase 3 LIBERTY ASTHMA TRAVERSE Trial. Allergy Asthma Immunol Res. 2024 Jul;16(4):372-386. doi: 10.4168/aair.2024.16.4.372. PMID 39155737
- [Derived] Maspero JF, Peters AT, Chapman KR, Domingo C, Stewart J, Hardin M, Maroni J, Tawo K, Khokhar FA, Mortensen E, Laws E, Radwan A, Jacob-Nara JA, Deniz Y, Rowe PJ. Long-Term Safety of Dupilumab in Patients With Moderate-to-Severe Asthma: TRAVERSE Continuation Study. J Allergy Clin Immunol Pract. 2024 Apr;12(4):991-997.e6. doi: 10.1016/j.jaip.2023.12.043. Epub 2023 Dec 30. PMID 38163585
- [Derived] Peters AT, Sagara H, Corren J, Domingo C, Altincatal A, Soler X, Pandit-Abid N, Crikelair N, Rowe PJ, Jacob-Nara JA, Deniz Y. Impact of dupilumab across seasons in patients with type 2, uncontrolled, moderate-to-severe asthma. Ann Allergy Asthma Immunol. 2024 Apr;132(4):477-484.e4. doi: 10.1016/j.anai.2023.11.021. Epub 2023 Nov 25. PMID 38013139
- [Derived] Wechsler ME, Souza-Machado A, Xu C, Mao X, Kapoor U, Khokhar FA, O'Malley JT, Petro CD, Casullo VM, Mannent LP, Rowe PJ, Jacob-Nara JA, Ruddy M, Laws E, Purcell LA, Hardin M. Preclinical and clinical experience with dupilumab on the correlates of live attenuated vaccines. J Allergy Clin Immunol Glob. 2021 Dec 8;1(1):9-15. doi: 10.1016/j.jacig.2021.12.003. eCollection 2022 Feb. PMID 37780074
- [Derived] Corren J, Hanania NA, Busse WW, Sher LD, Altincatal A, Hardin M, Mannent LP, Amin N, Lederer DJ, Soler X, Jacob-Nara JA, Rowe PJ, Deniz Y. Efficacy of dupilumab in patients with uncontrolled, moderate-to-severe asthma with fungal sensitization. Clin Exp Allergy. 2023 Oct;53(10):1020-1030. doi: 10.1111/cea.14389. Epub 2023 Sep 26. PMID 37752621
- [Derived] Pavord ID, Bourdin A, Papi A, Domingo C, Corren J, Altincatal A, Radwan A, Pandit-Abid N, Jacob-Nara JA, Deniz Y, Rowe PJ, Laws E, Lederer DJ, Hardin M. Dupilumab sustains efficacy in patients with moderate-to-severe type 2 asthma regardless of inhaled corticosteroids dose. Allergy. 2023 Nov;78(11):2921-2932. doi: 10.1111/all.15792. Epub 2023 Jul 11. PMID 37431558
- [Derived] Rabe KF, Pavord ID, Busse WW, Chupp GL, Izuhara K, Altincatal A, Gall R, Pandit-Abid N, Deniz Y, Rowe PJ, Jacob-Nara JA, Radwan A. Dupilumab improves long-term outcomes in patients with uncontrolled, moderate-to-severe GINA-based type 2 asthma, irrespective of allergic status. Allergy. 2023 Aug;78(8):2148-2156. doi: 10.1111/all.15747. Epub 2023 May 21. PMID 37073882
- [Derived] Sher LD, Corren J, Pavord ID, Daizadeh N, Altincatal A, Soler X, Djandji M, Radwan A, Jacob-Nara JA, Deniz Y, Rowe PJ. Dupilumab long-term efficacy in patients with non-OCS-dependent asthma with and without evidence of allergic asthma. J Asthma. 2023 Sep;60(9):1767-1774. doi: 10.1080/02770903.2023.2185895. Epub 2023 May 31. PMID 36876957
- [Derived] Sher LD, Passalacqua G, Taille C, Cohn L, Daizadeh N, Pandit-Abid N, Soler X, Khodzhayev A, Jacob-Nara JA, Deniz Y, Rowe PJ, Nag A, Zhang Y. The long-term effect of dupilumab on dyspnea, sleep, and activity in oral corticosteroid-dependent severe asthma. Ann Allergy Asthma Immunol. 2023 Mar;130(3):298-304. doi: 10.1016/j.anai.2022.12.002. Epub 2022 Dec 9. PMID 36509407
- [Derived] Berger P, Menzies-Gow A, Peters AT, Kuna P, Rabe KF, Altincatal A, Soler X, Pandit-Abid N, Siddiqui S, Jacob-Nara JA, Deniz Y, Rowe PJ. Long-term efficacy of dupilumab in asthma with or without chronic rhinosinusitis and nasal polyps. Ann Allergy Asthma Immunol. 2023 Feb;130(2):215-224. doi: 10.1016/j.anai.2022.11.006. Epub 2022 Nov 7. PMID 36356712
- [Derived] Tohda Y, Nakamura Y, Fujisawa T, Ebisawa M, Msihid J, Djandji M, Ortiz B, Jacob-Nara JA, Deniz Y, Rowe PJ, Ishida M, Arima K. Efficacy of dupilumab in patients with uncontrolled, moderate-to-severe asthma recruited from Japanese centers in the phase 3 LIBERTY ASTHMA TRAVERSE study. Allergol Int. 2023 Jan;72(1):89-99. doi: 10.1016/j.alit.2022.07.008. Epub 2022 Sep 13. PMID 36114102
- [Derived] Lugogo N, Mohan A. Are We Poised to Change the Trajectory of Maintenance Oral Corticosteroid Use in Severe Asthma in the Age of Biologics? Chest. 2022 Jul;162(1):4-5. doi: 10.1016/j.chest.2022.04.004. No abstract available. PMID 35809937
- [Derived] Wechsler ME, Klion AD, Paggiaro P, Nair P, Staumont-Salle D, Radwan A, Johnson RR, Kapoor U, Khokhar FA, Daizadeh N, Chen Z, Laws E, Ortiz B, Jacob-Nara JA, Mannent LP, Rowe PJ, Deniz Y. Effect of Dupilumab on Blood Eosinophil Counts in Patients With Asthma, Chronic Rhinosinusitis With Nasal Polyps, Atopic Dermatitis, or Eosinophilic Esophagitis. J Allergy Clin Immunol Pract. 2022 Oct;10(10):2695-2709. doi: 10.1016/j.jaip.2022.05.019. Epub 2022 May 28. PMID 35636689
- [Derived] Sher LD, Wechsler ME, Rabe KF, Maspero JF, Daizadeh N, Mao X, Ortiz B, Mannent LP, Laws E, Ruddy M, Pandit-Abid N, Jacob-Nara JA, Gall R, Rowe PJ, Deniz Y, Lederer DJ, Hardin M. Dupilumab Reduces Oral Corticosteroid Use in Patients With Corticosteroid-Dependent Severe Asthma: An Analysis of the Phase 3, Open-Label Extension TRAVERSE Trial. Chest. 2022 Jul;162(1):46-55. doi: 10.1016/j.chest.2022.01.071. Epub 2022 Feb 22. PMID 35217003
- [Derived] Wechsler ME, Ford LB, Maspero JF, Pavord ID, Papi A, Bourdin A, Watz H, Castro M, Nenasheva NM, Tohda Y, Langton D, Cardona G, Domingo C, Park HS, Chapman KR, Mao X, Zhang Y, Khan AH, Deniz Y, Rowe PJ, Kapoor U, Khokhar FA, Mannent LP, Ruddy M, Laws E, Amin N, Hardin M. Long-term safety and efficacy of dupilumab in patients with moderate-to-severe asthma (TRAVERSE): an open-label extension study. Lancet Respir Med. 2022 Jan;10(1):11-25. doi: 10.1016/S2213-2600(21)00322-2. Epub 2021 Sep 28. PMID 34597534

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was initiated at 365 sites in 27 countries. Participants who successfully completed treatment in studies DRI12544 (NCT01854047),EFC13579 (NCT02414854),EFC13691 (NCT02528214) and PDY14192 (NCT02573233) were eligible to continue their treatment in this extension study LTS12551. Total of 2282 participants were enrolled and treated in this study.
Pre-assignment Details: The Total study duration was maximum of 108 weeks for participants enrolled prior to amendment 4 approval and a maximum of 60 weeks for participants enrolled after amendment 4. Following amendment 4 (dated 31 Oct 2016) open-label treatment duration was amended to 48 weeks (1 year); and the 16-week post-treatment period was shortened to 12 weeks.
Groups:
- Participants From DRI12544: Placebo/Dupilumab: Participants who completed treatment of placebo (for dupilumab) and post-treatment period in study DRI12544, received a loading dose of dupilumab 600 milligram (mg) on Day 1 followed by a subcutaneous (SC) dose of dupilumab 300 mg every 2 weeks (q2w) for 96 weeks in combination with inhaled corticosteroid (ICS) therapy/long-acting beta-agonist (LABA) therapy in this extension study. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Participants From DRI12544: Dupilumab/Dupilumab: Participants who completed the treatment of dupilumab and post-treatment period in study DRI12544, received a loading dose of dupilumab 600 mg on Day 1 followed by a SC dose of dupilumab 300 mg q2w for 96 weeks in combination with ICS therapy/LABA therapy in this extension study. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Participants From EFC13579: Placebo/Dupilumab: Participants who completed the treatment of placebo (for dupilumab) in study EFC13579 and, who were enrolled before amendment 4 received a SC dose of dupilumab 300 mg q2w for 96 weeks and those who were enrolled after amendment 4 received a SC dose of dupilumab 300 mg q2w for 48 weeks in combination with ICS therapy/LABA therapy in this extension study. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Participants From EFC13579: Dupilumab/Dupilumab: Participants who completed the treatment for dupilumab in study EFC13579 and, who were enrolled before amendment 4 received a SC dose of dupilumab 300 mg q2w for 96 weeks and those who were enrolled after amendment 4 received a SC dose of dupilumab 300 mg q2w for 48 weeks in combination with ICS therapy/LABA therapy in this extension study. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Participants From EFC13691: Placebo/Dupilumab: Participants who completed the treatment of placebo (for dupilumab) in study EFC13691 and, who were enrolled before amendment 4 received a SC dose of dupilumab 300 mg q2w for 96 weeks and those who were enrolled after amendment 4 received a SC dose of dupilumab 300 mg q2w for 48 weeks in combination with oral corticosteroids (OCS) and ICS therapy in this extension study. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Participants From EFC13691: Dupilumab/Dupilumab: Participants who completed the treatment of dupilumab in study EFC13691 and, who were enrolled before amendment 4 received a SC dose of dupilumab 300 mg q2w for 96 weeks and those who were enrolled after amendment 4 received a SC dose of dupilumab 300 mg q2w for 48 weeks in combination with OCS and ICS therapy in this extension study. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Participants From PDY14192: Placebo/Dupilumab: Participants who completed the treatment of placebo (for dupilumab) in study PDY14192 received a SC dose of dupilumab 300 mg q2w for up to 96 weeks in combination with ICS therapy in this extension study. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Participants From PDY14192: Dupilumab/Dupilumab: Participants who completed the treatment of dupilumab in study PDY14192, received a SC dose of dupilumab 300 mg q2w for up to 96 weeks in combination with ICS therapy in this extension study. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
Period: Overall Study
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab | Participants From EFC13579: Placebo/Dupilumab | Participants From EFC13579: Dupilumab/Dupilumab | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab | Participants From PDY14192: Placebo/Dupilumab | Participants From PDY14192: Dupilumab/Dupilumab
Started (Participants who completed studies DRI12544, PDY14192, EFC13579, and EFC13691.) | 111 | 421 | 517 | 1013 | 97 | 90 | 19 | 14
Completed | 102 | 379 | 465 | 908 | 83 | 76 | 15 | 11
Not Completed | 9 | 42 | 52 | 105 | 14 | 14 | 4 | 3
Not completed — Lack of Efficacy | 1 | 0 | 3 | 2 | 1 | 2 | 1 | 0
Not completed — Poor compliance to protocol | 1 | 1 | 3 | 7 | 1 | 1 | 0 | 0
Not completed — Other unspecified | 4 | 22 | 33 | 64 | 8 | 6 | 2 | 1
Not completed — Adverse Event | 3 | 19 | 13 | 32 | 4 | 5 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled participants.
Groups:
- Participants From DRI12544: Placebo/Dupilumab: Participants who completed treatment of placebo (for dupilumab) and post-treatment period in study DRI12544, received a loading dose of dupilumab 600 mg on Day 1 followed by a SC dose of dupilumab 300 mg q2w for 96 weeks in combination with ICS therapy/LABA therapy in this extension study. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Participants From EFC13691: Placebo/Dupilumab: Participants who completed the treatment of placebo (for dupilumab) in study EFC13691 and, who were enrolled before amendment 4 received a SC dose of dupilumab 300 mg q2w for 96 weeks and those who were enrolled after amendment 4 received a SC dose of dupilumab 300 mg q2w for 48 weeks in combination with OCS and ICS therapy in this extension study. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Total: Total of all reporting groups
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab | Participants From EFC13579: Placebo/Dupilumab | Participants From EFC13579: Dupilumab/Dupilumab | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab | Participants From PDY14192: Placebo/Dupilumab | Participants From PDY14192: Dupilumab/Dupilumab | Total
Number analyzed (Participants) | 111 | 421 | 517 | 1013 | 97 | 90 | 19 | 14 | 2282
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 32 | 55 | 1 | 1 | 0 | 0 | 89
  18-64 years | 101 | 374 | 422 | 826 | 81 | 80 | 19 | 14 | 1917
  65-74 years | 8 | 40 | 59 | 112 | 14 | 8 | 0 | 0 | 241
  75-84 years | 2 | 7 | 4 | 20 | 1 | 1 | 0 | 0 | 35
  ≥85 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 259 | 335 | 618 | 57 | 53 | 7 | 10 | 1408
  Male | 42 | 162 | 182 | 395 | 40 | 37 | 12 | 4 | 874
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Asian | 18 | 70 | 51 | 116 | 1 | 0 | 0 | 1 | 257
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3
  Black or African American | 1 | 8 | 17 | 43 | 1 | 2 | 2 | 1 | 75
  White | 88 | 339 | 445 | 844 | 91 | 86 | 17 | 12 | 1922
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 4 | 9 | 2 | 1 | 0 | 0 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which did not necessarily had to have causal relationship with treatment. TEAEs were defined as AEs that developed, worsened, or became serious during the treatment emergent AE period (time from first dose of investigational medicinal product [IMP] in LTS12551 up to the last dose of dupilumab plus 14 weeks). A Serious AE (SAE) was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event.
Time Frame: From the first IMP injection in LTS12551 to the last IMP injection plus 14 weeks (up to 108 weeks)
Population: Analysis was performed on exposed population which included participants who actually received at least 1 dose or part of a dose of the IMP in LTS12551 study.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab | Participants From EFC13579: Placebo/Dupilumab | Participants From EFC13579: Dupilumab/Dupilumab | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab | Participants From PDY14192: Placebo/Dupilumab | Participants From PDY14192: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421 | 517 | 1013 | 97 | 90 | 19 | 14
Participants
  Any TEAE | 88 | 369 | 414 | 789 | 74 | 70 | 18 | 13
  Any treatment emergent SAE | 14 | 42 | 48 | 106 | 12 | 10 | 0 | 4
  Any TEAE leading to death | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0
  Any TEAE leading to permanent discontinuation | 3 | 19 | 12 | 31 | 4 | 5 | 1 | 2

2. Secondary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Abnormalities During the TEAE Period
Description: Criteria for potentially clinically significant vital sign abnormalities:
  * Systolic blood pressure (SBP): Less than or equal to (≤) 95 Adults (≤90 Adolescents) millimeters of mercury (mmHg) and decrease from baseline (DFB) greater than or equal to (≥) 20 mmHg; ≥ 160 Adults (≥ 119 Adolescents) mmHg and increase from baseline (IFB) ≥ 20 mmHg.
  * Diastolic blood pressure (DBP): ≤ 45 Adults (≤54 Adolescents) mmHg and DFB ≥ 10 mmHg; ≥ 110 Adults (≥78 Adolescents) mmHg and IFB ≥ 10 mmHg.
  * Heart rate (HR): ≤ 50 beats per minute (bpm) and DFB ≥ 20 bpm; ≥ 120 bpm and IFB ≥ 20 bpm.
  * Respiratory rate: less than (<) 12 breaths/min(b/m); greater than (>) 20 b/m.
  * Weight (kg): ≥ 5 percent (%) DFB; ≥ 5% IFB.
  * Temperature: ≥ 38.0 degree Celsius (°C) rectal/ear/temporal; ≥ 37.5°C oral; ≥ 37.2°C axillary.
  TEAE period was defined as the time from first dose of IMP in LTS12551 up to the last dose of dupilumab plus 14 weeks.
Time Frame: From the first IMP injection in LTS12551 to the last IMP injection plus 14 weeks (up to 108 weeks)
Population: Analysis was performed on exposed population. Here, 'number analyzed' = number of participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab | Participants From EFC13579: Placebo/Dupilumab | Participants From EFC13579: Dupilumab/Dupilumab | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab | Participants From PDY14192: Placebo/Dupilumab | Participants From PDY14192: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421 | 517 | 1013 | 97 | 90 | 19 | 14
Participants
  SBP: ≤ 95 (≤90) & DFB ≥ 20 mmHg: number analyzed (Participants) | 111 | 421 | 516 | 1013 | 97 | 90 | 19 | 14
  SBP: ≤ 95 (≤90) & DFB ≥ 20 mmHg | 4 | 12 | 19 | 40 | 0 | 1 | 2 | 0
  SBP: ≥ 160 (≥119) & IFB ≥ 20 mmHg: number analyzed (Participants) | 111 | 421 | 516 | 1013 | 97 | 90 | 19 | 14
  SBP: ≥ 160 (≥119) & IFB ≥ 20 mmHg | 2 | 17 | 21 | 45 | 6 | 1 | 1 | 3
  DBP: ≤ 45 (≤54) & DFB ≥ 10 mmHg: number analyzed (Participants) | 111 | 421 | 516 | 1013 | 97 | 90 | 19 | 14
  DBP: ≤ 45 (≤54) & DFB ≥ 10 mmHg | 1 | 1 | 11 | 15 | 0 | 0 | 0 | 0
  DBP: ≥ 110 (≥78) & IFB ≥ 10 mmHg: number analyzed (Participants) | 111 | 421 | 516 | 1013 | 97 | 90 | 19 | 14
  DBP: ≥ 110 (≥78) & IFB ≥ 10 mmHg | 0 | 4 | 15 | 20 | 2 | 0 | 0 | 0
  HR: ≤ 50 & DFB ≥ 20 bpm: number analyzed (Participants) | 111 | 421 | 516 | 1013 | 97 | 90 | 19 | 14
  HR: ≤ 50 & DFB ≥ 20 bpm | 0 | 3 | 2 | 12 | 0 | 0 | 0 | 0
  HR: ≥ 120 & IFB ≥ 20 bpm: number analyzed (Participants) | 111 | 421 | 516 | 1013 | 97 | 90 | 19 | 14
  HR: ≥ 120 & IFB ≥ 20 bpm | 0 | 0 | 2 | 5 | 1 | 0 | 0 | 0
  Respiratory rate: < 12 b/m: number analyzed (Participants) | 111 | 421 | 516 | 1013 | 97 | 90 | 19 | 14
  Respiratory rate: < 12 b/m | 5 | 17 | 18 | 24 | 4 | 0 | 2 | 3
  Respiratory rate: > 20 b/m: number analyzed (Participants) | 111 | 421 | 516 | 1013 | 97 | 90 | 19 | 14
  Respiratory rate: > 20 b/m | 23 | 104 | 88 | 195 | 18 | 12 | 4 | 0
  Weight: ≥ 5% DFB: number analyzed (Participants) | 111 | 421 | 516 | 1013 | 97 | 90 | 19 | 14
  Weight: ≥ 5% DFB | 32 | 106 | 146 | 261 | 22 | 29 | 3 | 3
  Weight: ≥ 5% IFB: number analyzed (Participants) | 111 | 421 | 485 | 958 | 96 | 89 | 19 | 14
  Weight: ≥ 5% IFB | 45 | 181 | 189 | 378 | 29 | 37 | 8 | 5
  Temperature: ≥ 38.0°C: number analyzed (Participants) | 111 | 421 | 516 | 1013 | 97 | 90 | 19 | 14
  Temperature: ≥ 38.0°C | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Temperature: ≥ 37.5°C: number analyzed (Participants) | 111 | 421 | 516 | 1013 | 97 | 90 | 19 | 14
  Temperature: ≥ 37.5°C | 1 | 0 | 9 | 6 | 0 | 0 | 0 | 0
  Temperature: ≥ 37.2°C: number analyzed (Participants) | 111 | 421 | 516 | 1013 | 97 | 90 | 19 | 14
  Temperature: ≥ 37.2°C | 3 | 21 | 4 | 16 | 0 | 1 | 0 | 0

3. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Hematological Parameters (Red Blood Cells [RBCs], Platelets and Coagulation) During the TEAE Period
Description: Criteria for potentially clinically significant abnormalities:
  * Hemoglobin (Hb): ≤ 115 grams per liter (g/L)(Male [M]), ≤ 95 g/L (Female[ F]) (< 100 g/L Adolescents); ≥ 185 g/L (M), ≥ 165 g/L (F) (≥ 200 g/L Adolescents); DFB ≥ 20 g/L.
  * Hematocrit: ≤ 0.37 volume/volume (v/v) (M); ≤ 0.32 v/v (F) (<0.32 v/v Adolescents); ≥ 0.55 v/v (M); 0.5 v/v (F) (>0.47 v/v Adolescents).
  * RBCs: ≥ 6 Tera/L.
  * Platelets: < 100 Giga(G)/L; ≥ 700 G/L.
  TEAE period was defined as the time from first dose of IMP in LTS12551 up to the last dose of dupilumab plus 14 weeks.
Time Frame: From the first IMP injection in LTS12551 to the last IMP injection plus 14 weeks (up to 108 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab | Participants From EFC13579: Placebo/Dupilumab | Participants From EFC13579: Dupilumab/Dupilumab | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab | Participants From PDY14192: Placebo/Dupilumab | Participants From PDY14192: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421 | 517 | 1013 | 97 | 90 | 19 | 14
Participants
  Hb: ≤ 115 g/L, ≤ 95 g/L (< 100 g/L): number analyzed (Participants) | 111 | 421 | 514 | 1009 | 97 | 90 | 19 | 14
  Hb: ≤ 115 g/L, ≤ 95 g/L (< 100 g/L) | 2 | 7 | 12 | 29 | 0 | 3 | 0 | 0
  Hb: ≥ 185 g/L, ≥ 165 g/L(≥ 200 g/L): number analyzed (Participants) | 111 | 421 | 514 | 1009 | 97 | 90 | 19 | 14
  Hb: ≥ 185 g/L, ≥ 165 g/L(≥ 200 g/L) | 1 | 3 | 8 | 4 | 2 | 1 | 0 | 0
  Hb: DFB ≥ 20 g/L: number analyzed (Participants) | 111 | 421 | 513 | 1008 | 97 | 90 | 19 | 14
  Hb: DFB ≥ 20 g/L | 13 | 41 | 40 | 118 | 11 | 7 | 0 | 0
  Hematocrit: ≤ 0.37 v/v; ≤ 0.32 v/v(<0.32 v/v): number analyzed (Participants) | 111 | 421 | 514 | 1007 | 97 | 90 | 19 | 14
  Hematocrit: ≤ 0.37 v/v; ≤ 0.32 v/v(<0.32 v/v) | 6 | 19 | 23 | 47 | 3 | 5 | 0 | 0
  Hematocrit: ≥ 0.55 v/v; ≥ 0.5 v/v(>0.47 v/v): number analyzed (Participants) | 111 | 421 | 514 | 1007 | 97 | 90 | 19 | 14
  Hematocrit: ≥ 0.55 v/v; ≥ 0.5 v/v(>0.47 v/v) | 3 | 6 | 26 | 36 | 3 | 3 | 0 | 0
  RBCs: ≥ 6 Tera/L: number analyzed (Participants) | 111 | 421 | 514 | 1009 | 97 | 90 | 19 | 14
  RBCs: ≥ 6 Tera/L | 1 | 5 | 8 | 15 | 0 | 2 | 0 | 1
  Platelets: < 100G/ L: number analyzed (Participants) | 111 | 421 | 514 | 1007 | 97 | 90 | 19 | 14
  Platelets: < 100G/ L | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 1
  Platelets: ≥ 700 G/L: number analyzed (Participants) | 111 | 421 | 514 | 1007 | 97 | 90 | 19 | 14
  Platelets: ≥ 700 G/L | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Severe Exacerbation Events
Description: Severe asthma exacerbation events were defined as a deterioration of asthma which required: use of systemic corticosteroids for ≥ 3 days, (participants from study EFC13691 (NCT02528214), and who were taking systemic corticosteroids: the use of systemic corticosteroids at least double the current dose and for ≥3 days.) or, hospitalization or emergency room visit because of asthma, required systemic corticosteroids.
Time Frame: From the first IMP injection in LTS12551 to the last IMP injection plus 2 weeks (up to 96 weeks)
Population: Analysis was performed on exposed population.
Measure: Number; unit: number of events
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab | Participants From EFC13579: Placebo/Dupilumab | Participants From EFC13579: Dupilumab/Dupilumab | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab | Participants From PDY14192: Placebo/Dupilumab | Participants From PDY14192: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421 | 517 | 1013 | 97 | 90 | 19 | 14
number of events | 62 | 242 | 234 | 437 | 35 | 41 | 3 | 1

5. Secondary Outcome: Annualized Event Rate Per Participant-Years for Severe Exacerbation
Description: The annualized event rate per participant-years was defined as the total number of events that occurred during the treatment period divided by the total number of participant-years during the treatment period.
Time Frame: From the first IMP injection in LTS12551 to the last IMP injection plus 2 weeks (up to 96 weeks)
Population: Analysis was performed on exposed population.
Measure: Number; unit: exacerbation per participant-years
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab | Participants From EFC13579: Placebo/Dupilumab | Participants From EFC13579: Dupilumab/Dupilumab | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab | Participants From PDY14192: Placebo/Dupilumab | Participants From PDY14192: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421 | 517 | 1013 | 97 | 90 | 19 | 14
exacerbation per participant-years | 0.314 | 0.330 | 0.351 | 0.331 | 0.302 | 0.391 | 0.149 | 0.077

6. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Weeks 48 and 96
Description: FEV1 was the volume of air exhaled from the lungs in the first second of a forced expiration as measured by spirometer. For this analysis, baseline was defined as respective parent study baseline.
Time Frame: Baseline of parent study, Week 48 and Week 96 of this extension study
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab | Participants From EFC13579: Placebo/Dupilumab | Participants From EFC13579: Dupilumab/Dupilumab | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab | Participants From PDY14192: Placebo/Dupilumab | Participants From PDY14192: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421 | 517 | 1013 | 97 | 90 | 19 | 14
liters
  Week 48: number analyzed (Participants) | 105 | 396 | 486 | 951 | 88 | 82 | 16 | 11
  Week 48 | 0.24 (0.42) | 0.28 (0.45) | 0.34 (0.44) | 0.36 (0.53) | 0.31 (0.50) | 0.33 (0.53) | 0.23 (0.40) | 0.01 (0.21)
  Week 96: number analyzed (Participants) | 102 | 380 | 219 | 447 | 32 | 28 | 5 | 2
  Week 96 | 0.22 (0.44) | 0.27 (0.46) | 0.33 (0.44) | 0.31 (0.47) | 0.36 (0.66) | 0.25 (0.46) | 0.14 (0.41) | 0.01 (0.12)

7. Secondary Outcome: Change From Baseline in Percent Predicted FEV1 at Weeks 48 and 96
Description: as for outcome 6
Time Frame: Baseline of parent study, Week 48 and Week 96 of this extension study
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent predicted FEV1
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab | Participants From EFC13579: Placebo/Dupilumab | Participants From EFC13579: Dupilumab/Dupilumab | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab | Participants From PDY14192: Placebo/Dupilumab | Participants From PDY14192: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421 | 517 | 1013 | 97 | 90 | 19 | 14
percent predicted FEV1
  Week 48: number analyzed (Participants) | 105 | 396 | 486 | 951 | 88 | 82 | 16 | 11
  Week 48 | 9.21 (13.61) | 10.42 (14.61) | 11.74 (14.27) | 12.16 (16.58) | 10.45 (15.03) | 12.41 (18.27) | 5.88 (10.06) | 1.36 (8.35)
  Week 96: number analyzed (Participants) | 102 | 380 | 219 | 447 | 32 | 28 | 5 | 2
  Week 96 | 8.86 (14.47) | 10.68 (15.10) | 12.53 (14.50) | 11.25 (14.55) | 13.06 (19.57) | 10.00 (15.79) | 4.20 (9.60) | 2.00 (2.83)

8. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Weeks 48 and 96
Description: FVC was a standard pulmonary function test used to quantify respiratory muscle weakness. FVC was the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. For this analysis, baseline was defined as respective parent study baseline.
Time Frame: Baseline of parent study, Week 48, and Week 96 of this extension study
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab | Participants From EFC13579: Placebo/Dupilumab | Participants From EFC13579: Dupilumab/Dupilumab | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab | Participants From PDY14192: Placebo/Dupilumab | Participants From PDY14192: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421 | 517 | 1013 | 97 | 90 | 19 | 14
liters
  Week 48: number analyzed (Participants) | 105 | 396 | 486 | 951 | 88 | 82 | 16 | 11
  Week 48 | 0.22 (0.45) | 0.25 (0.50) | 0.30 (0.48) | 0.35 (0.60) | 0.29 (0.56) | 0.38 (0.56) | 0.21 (0.42) | 0.05 (0.30)
  Week 96: number analyzed (Participants) | 102 | 380 | 219 | 447 | 32 | 28 | 5 | 2
  Week 96 | 0.16 (0.47) | 0.22 (0.52) | 0.27 (0.48) | 0.25 (0.50) | 0.38 (0.82) | 0.22 (0.42) | 0.08 (0.29) | 0.05 (0.40)

9. Secondary Outcome: Change From Baseline in Forced Expiratory Flow (FEF) 25-75% at Weeks 48 and 96
Description: FEF was the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. FEF 25-75% was defined as the mean FEF between 25% and 75% of the FVC, where FVC was defined as the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. For this analysis, baseline was defined as respective parent study baseline.
Time Frame: Baseline of parent study, Week 48, and Week 96 of this extension study
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liters/second
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab | Participants From EFC13579: Placebo/Dupilumab | Participants From EFC13579: Dupilumab/Dupilumab | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab | Participants From PDY14192: Placebo/Dupilumab | Participants From PDY14192: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421 | 517 | 1013 | 97 | 90 | 19 | 14
liters/second
  Week 48: number analyzed (Participants) | 105 | 396 | 486 | 951 | 88 | 82 | 16 | 11
  Week 48 | 0.27 (0.55) | 0.31 (0.55) | 0.39 (0.57) | 0.39 (0.66) | 0.34 (0.56) | 0.29 (0.66) | 0.23 (0.44) | 0.04 (0.26)
  Week 96: number analyzed (Participants) | 102 | 380 | 219 | 447 | 32 | 28 | 5 | 2
  Week 96 | 0.28 (0.57) | 0.32 (0.55) | 0.38 (0.53) | 0.36 (0.61) | 0.42 (0.64) | 0.27 (0.53) | 0.19 (0.41) | 0.04 (0.14)

10. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire 5-Question Version (ACQ-5) Mean Scores at Weeks 24 and 48
Description: The ACQ-5 had 5 questions, reflecting the top-scoring five asthma symptoms: woken at night by symptoms, wake in the mornings with symptoms, limitation of daily activities, shortness of breath and wheeze. Participants were asked to recall how their asthma had been during the previous week and to respond to each of the five symptom questions on a 7-point scale ranged from 0 (no impairment) to 6 (maximum impairment). ACQ-5 total mean score was mean of the scores of all 5 questions and, therefore, ranged from 0 (totally controlled) to 6 (severely uncontrolled), higher scores indicated lower asthma control. For this analysis, baseline was defined as respective parent study baseline.
Time Frame: Baseline of parent study, Weeks 24, and 48 of this extension study
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab | Participants From EFC13579: Placebo/Dupilumab | Participants From EFC13579: Dupilumab/Dupilumab | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab | Participants From PDY14192: Placebo/Dupilumab | Participants From PDY14192: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421 | 517 | 1013 | 97 | 90 | 19 | 14
score on a scale
  Week 24: number analyzed (Participants) | 110 | 421 | 513 | 1005 | 96 | 87 | 19 | 13
  Week 24 | -1.37 (0.91) | -1.48 (1.10) | -1.61 (1.08) | -1.68 (1.05) | -1.09 (1.10) | -1.15 (1.17) | -0.96 (1.03) | -0.80 (0.46)
  Week 48: number analyzed (Participants) | 105 | 400 | 488 | 957 | 90 | 78 | 15 | 11
  Week 48 | -1.33 (1.07) | -1.57 (1.11) | -1.64 (1.08) | -1.69 (1.08) | -1.21 (1.00) | -1.06 (1.25) | -0.89 (1.02) | -0.87 (0.58)

11. Secondary Outcome: Percentage of Participants Achieving ACQ-5 Score Response (ACQ-5 Responders) at Weeks 24 and 48
Description: ACQ-5 response was defined as change from baseline in ACQ-5 scores ≥ 0.5. The ACQ-5 had 5 questions, reflecting the top-scoring five asthma symptoms: woken at night by symptoms, wake in the mornings with symptoms, limitation of daily activities, shortness of breath and wheeze. Participants were asked to recall how their asthma had been during the previous week and to respond to each of the five symptom questions on a 7-point scale ranged from 0 (no impairment) to 6 (maximum impairment). ACQ-5 mean total score was mean of the scores of all 5 questions and, therefore, ranged from 0 (totally controlled) to 6 (severely uncontrolled). Higher score indicated lower asthma control.
Time Frame: At Weeks 24, and 48 of this extension study
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab | Participants From EFC13579: Placebo/Dupilumab | Participants From EFC13579: Dupilumab/Dupilumab | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab | Participants From PDY14192: Placebo/Dupilumab | Participants From PDY14192: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421 | 517 | 1013 | 97 | 90 | 19 | 14
percentage of participants
  Week 24: number analyzed (Participants) | 110 | 421 | 513 | 1005 | 96 | 87 | 19 | 13
  Week 24 | 82.7 | 80.8 | 84.0 | 86.5 | 67.7 | 70.1 | 57.9 | 69.2
  Week 48: number analyzed (Participants) | 105 | 400 | 488 | 957 | 90 | 78 | 15 | 11
  Week 48 | 79.0 | 82.3 | 85.7 | 86.7 | 75.6 | 70.5 | 60.0 | 72.7

12. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire (AQLQ) Global Scores at Weeks 24 and 48
Description: The AQLQ was designed to measure the functional impairments that are most troublesome to adults as a result of their asthma. The AQLQ comprised of 32 items in 4 domains: symptoms (12 items), activity limitation (11 items), emotional function (5 items), and environmental stimuli (4 items). Each item was scored on a 7-point likert scale ranged from 1=severely impaired to 7=not impaired. The 32 items of the questionnaire were averaged to produce one overall quality of life score ranging from 1 (severely impaired) to 7 (not impaired); higher scores indicated better quality of life. For this analysis, baseline was defined as respective parent study baseline.
Time Frame: Baseline of parent study, Weeks 24, and 48 of this extension study
Population: Analysis was performed on exposed population. Here, 'number analyzed' = number of participants with available data for each specified category. Data were planned to be collected and analyzed for the participants from Studies DRI12544, EFC13579, and EFC13691 only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab | Participants From EFC13579: Placebo/Dupilumab | Participants From EFC13579: Dupilumab/Dupilumab | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421 | 517 | 1013 | 97 | 90
score on a scale
  Week 24: number analyzed (Participants) | 108 | 413 | 495 | 948 | 95 | 88
  Week 24 | 1.07 (0.99) | 1.28 (1.24) | 1.38 (1.15) | 1.38 (1.16) | 0.99 (1.10) | 0.97 (1.26)
  Week 48: number analyzed (Participants) | 103 | 397 | 473 | 908 | 90 | 79
  Week 48 | 1.07 (1.13) | 1.40 (1.19) | 1.39 (1.17) | 1.40 (1.18) | 1.06 (0.98) | 1.00 (1.23)

13. Secondary Outcome: Percentage of Participants Achieving AQLQ Global Score Response (AQLQ Responders) at Weeks 24 and 48
Description: AQLQ global response was defined as participants with change from baseline in AQLQ global score ≥ 0.5. The AQLQ was designed to measure the functional impairments that are most troublesome to adults as a result of their asthma. The AQLQ comprised of 32 items in 4 domains: symptoms (12 items), activity limitation (11 items), emotional function (5 items), environmental stimuli (4 items). Each item was scored on a 7-point likert scale (1=severely impaired, 7=not impaired). The 32 items of the questionnaire are averaged to produce one overall quality of life score ranging from 1 (severely impaired) to 7 (not impaired). Higher scores indicated better quality of life.
Time Frame: At Weeks 24, and 48 of this extension study
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab | Participants From EFC13579: Placebo/Dupilumab | Participants From EFC13579: Dupilumab/Dupilumab | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421 | 517 | 1013 | 97 | 90
percentage of participants
  Week 24: number analyzed (Participants) | 108 | 413 | 495 | 948 | 95 | 88
  Week 24 | 67.6 | 73.6 | 77.6 | 77.2 | 64.2 | 61.4
  Week 48: number analyzed (Participants) | 103 | 397 | 473 | 908 | 90 | 79
  Week 48 | 65.0 | 76.3 | 77.4 | 78.4 | 73.3 | 68.4

14. Secondary Outcome: Serum Concentrations of Dupilumab Over Time Till Week 96
Description: For this analysis, baseline was defined as respective parent study baseline. Here, 'number analyzed'=number of participants with available data for each specified category.
Time Frame: Baseline of parent study, Weeks 0, 4, 12, 24, 48, 72, and 96 of this extension study
Population: Analysis was performed on Pharmacokinetics (PK) population which consisted of all the participants who had actually received at least one dose or part of a dose of dupilumab in the LTS12551 study, with at least one non-missing and evaluable pre-dose serum concentration value after the first dose of dupilumab in the LTS12551 study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab | Participants From EFC13579: Placebo/Dupilumab | Participants From EFC13579: Dupilumab/Dupilumab | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab | Participants From PDY14192: Placebo/Dupilumab | Participants From PDY14192: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421 | 515 | 1008 | 96 | 90 | 19 | 14
nanogram per milliliter (ng/mL)
  Baseline: number analyzed (Participants) | 110 | 413 | 0 | 993 | 0 | 88 | 0 | 14
  Baseline | 0.00 (0.000) | 0.00 (1990.640) |  | 0.00 (2286.888) |  | 0.00 (0.000) |  | 0.00 (0.000)
  Week 0: number analyzed (Participants) | 110 | 417 | 0 | 968 | 0 | 88 | 0 | 14
  Week 0 | 0.00 (0.000) | 0.00 (0.000) |  | 37230.97 (73.261) |  | 40754.49 (54.858) |  | 52545.41 (44.678)
  Week 4: number analyzed (Participants) | 109 | 414 | 500 | 971 | 93 | 88 | 18 | 13
  Week 4 | 46848.70 (43.149) | 40704.77 (47.293) | 25847.86 (49.371) | 50566.66 (55.104) | 25868.25 (53.450) | 48295.93 (52.655) | 23336.89 (50.542) | 56486.58 (45.755)
  Week 12: number analyzed (Participants) | 111 | 417 | 501 | 973 | 94 | 87 | 16 | 12
  Week 12 | 54467.13 (50.267) | 48155.26 (52.353) | 45406.55 (51.399) | 55140.49 (53.114) | 44064.95 (57.100) | 50904.34 (51.233) | 49026.51 (41.619) | 55365.35 (53.317)
  Week 24: number analyzed (Participants) | 108 | 405 | 500 | 973 | 90 | 83 | 16 | 11
  Week 24 | 47023.84 (51.645) | 49730.56 (53.625) | 50984.57 (53.744) | 54897.58 (54.044) | 57363.72 (57.889) | 44219.42 (55.383) | 63080.82 (51.224) | 60643.16 (41.617)
  Week 48: number analyzed (Participants) | 106 | 397 | 484 | 951 | 89 | 82 | 16 | 11
  Week 48 | 46355.26 (52.612) | 45919.75 (55.932) | 41867.50 (60.345) | 41849.96 (62.049) | 36219.47 (67.530) | 36564.41 (60.959) | 24864.79 (58.016) | 53320.11 (46.714)
  Week 72: number analyzed (Participants) | 105 | 385 | 227 | 453 | 35 | 29 | 5 | 2
  Week 72 | 44771.52 (56.256) | 46842.64 (53.335) | 45628.10 (56.232) | 46372.55 (57.719) | 60117.76 (62.390) | 32029.19 (66.785) | 40362.88 (55.567) | 26383.90 (120.013)
  Week 96: number analyzed (Participants) | 101 | 381 | 222 | 446 | 33 | 29 | 5 | 2
  Week 96 | 42431.08 (59.222) | 42661.18 (59.658) | 38908.58 (64.633) | 39088.60 (62.897) | 49810.65 (65.546) | 19030.70 (67.237) | 42360.37 (49.409) | 56378.01 (7.140)

15. Secondary Outcome: Percentage of Participants With Antidrug Antibodies (ADA) Response
Description: ADA response were categorized as: treatment emergent and treatment boosted response. 1) Treatment emergent was defined as an ADA positive response in the assay post first dose in LTS12551, when baseline results were negative or missing. 2) Treatment boosted was defined as: an ADA positive response in the assay post first dose that was greater-than or equal to 4-fold over baseline titer levels, when baseline results were positive. The criteria for positive was defined as "30 to > 10,000", where low titer (< 1,000); moderate (1,000 ≤ titer ≤ 10,000) and high titer (> 10,000).
Time Frame: From the first IMP injection in LTS12551 to the last IMP injection plus 2 weeks (up to 96 weeks)
Population: Analysis was performed on ADA population which consisted of all participants who had actually received at least one dose or part of a dose of dupilumab in the LTS12551 study, with at least one pre-dose sample that was assayed successfully using the ADA assay after the first dose of dupilumab in the LTS12551 study.
Measure: Number; unit: percentage of participants
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab | Participants From EFC13579: Placebo/Dupilumab | Participants From EFC13579: Dupilumab/Dupilumab | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab | Participants From PDY14192: Placebo/Dupilumab | Participants From PDY14192: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421 | 515 | 1008 | 95 | 90 | 19 | 14
percentage of participants
  Treatment-emergent ADA | 10.8 | 12.1 | 9.5 | 4.5 | 7.4 | 8.9 | 0 | 7.1
  Treatment-boosted ADA | 0 | 0 | 0 | 0 | 1.1 | 0 | 0 | 0

16. Secondary Outcome: Change From Baseline in Blood Eosinophils Cells Count at Weeks 48 and 96
Description: For this analysis, baseline was defined as respective parent study baseline.
Time Frame: Baseline of parent study, Week 48 and Week 96 of this extension study
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab | Participants From EFC13579: Placebo/Dupilumab | Participants From EFC13579: Dupilumab/Dupilumab | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab | Participants From PDY14192: Placebo/Dupilumab | Participants From PDY14192: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421 | 517 | 1013 | 97 | 90 | 19 | 14
10^9 cells/L
  Week 48: number analyzed (Participants) | 103 | 386 | 474 | 935 | 87 | 82 | 14 | 10
  Week 48 | 0.007 (0.475) | -0.041 (0.588) | -0.096 (0.428) | -0.099 (0.360) | 0.098 (0.450) | 0.016 (0.382) | -0.066 (0.181) | -0.026 (0.187)
  Week 96: number analyzed (Participants) | 102 | 381 | 218 | 435 | 30 | 29 | 4 | 2
  Week 96 | -0.074 (0.251) | -0.081 (0.562) | -0.161 (0.391) | -0.114 (0.354) | -0.051 (0.399) | 0.083 (0.642) | -0.103 (0.039) | 0.025 (0.134)

17. Secondary Outcome: Change From Baseline in Morning Peak Expiratory Flow (PEF) at Weeks 48 and 96: Participants From Study DRI12544
Description: The PEF was a participant's maximum speed of expiration, as measured with a peak flow meter. Peak flow testing for PEF was performed at morning and evening. Morning PEF was performed within 15 minutes after arising (between 5:30 AM and 10 AM) prior to taking any salbutamol/albuterol or levosalbutamol/levalbuterol. For this analysis, baseline was defined as parent study DRI12544 baseline.
Time Frame: Baseline of parent study, Week 48 and Week 96 of this extension study
Population: Analysis was performed on exposed population. Here, 'number analyzed' = number of participants with available data for each specified category. Data were planned to be collected and analyzed only for the participants from Study DRI12544 and not for the participants from other studies.
Measure: Mean (Standard Deviation); unit: liters per minute (L/min)
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421
liters per minute (L/min)
  Week 48: number analyzed (Participants) | 110 | 407
  Week 48 | 13.26 (76.71) | 22.95 (70.06)
  Week 96: number analyzed (Participants) | 92 | 340
  Week 96 | 13.63 (83.88) | 21.69 (77.70)

18. Secondary Outcome: Change From Baseline in Evening Peak Expiratory Flow (PEF) at Weeks 48 and 96: Participants From Study DRI12544
Description: The PEF was a participant's maximum speed of expiration, as measured with a peak flow meter. Peak flow testing for PEF was performed at morning and evening. Evening PEF was performed in the evening (between 5:30 PM and 10 PM) prior to taking any salbutamol/albuterol or levosalbutamol/levalbuterol. For this analysis, baseline was defined as parent DRI12544 study baseline.
Time Frame: Baseline of parent study, Week 48 and Week 96 of this extension study
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421
L/min
  Week 48: number analyzed (Participants) | 109 | 406
  Week 48 | 4.65 (75.00) | 11.97 (72.19)
  Week 96: number analyzed (Participants) | 89 | 327
  Week 96 | 1.16 (79.47) | 10.05 (79.47)

19. Secondary Outcome: Change From Baseline in Morning Asthma Symptom Scores at Weeks 48 and 96: Participants From Study DRI12544
Description: Morning asthma symptom score was determined using AM (ante meridiem) symptom scoring system which evaluated participant's overall asthma symptoms experienced during the night. It ranges from 0 to 4 as: 0=no asthma symptoms, slept through the night, 1=slept well, but some complaints in the morning. No nighttime awakenings, 2=woke up once because of asthma (including early awakening), 3=woke up several times because of asthma (including early awakening), 4=bad night, awake most of the night because of asthma; higher scores indicated more severe symptoms. For this analysis, baseline was defined as parent DRI12544 study baseline.
Time Frame: Baseline of parent study, Week 48 and Week 96 of this extension study
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421
score on a scale
  Week 48: number analyzed (Participants) | 110 | 410
  Week 48 | -0.49 (0.78) | -0.68 (0.79)
  Week 96: number analyzed (Participants) | 92 | 324
  Week 96 | -0.52 (0.90) | -0.76 (0.81)

20. Secondary Outcome: Change From Baseline in Evening Asthma Symptom Scores at Weeks 48 and 96: Participants From Study DRI12544
Description: Evening asthma symptom score was determined using PM (post meridiem) symptom scoring system which evaluated participant's overall asthma symptoms experienced during the day. It ranged from 0 to 4 as: 0=very well, no asthma symptoms, 1=one episode of wheezing, cough, or breathlessness, 2=more than one episode of wheezing, cough, or breathlessness without interference of normal activities, 3=wheezing, cough, or breathlessness most of the day, which interfered to some extent with normal activities, 4=asthma very bad, unable to carry out daily activities as usual; higher scores indicated more severe symptoms. For this analysis, baseline was defined as parent DRI12544 study baseline.
Time Frame: Baseline of parent study, Week 48, and Week 96 of this extension study
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421
score on a scale
  Week 48: number analyzed (Participants) | 109 | 407
  Week 48 | -0.47 (0.81) | -0.72 (0.85)
  Week 96: number analyzed (Participants) | 88 | 330
  Week 96 | -0.49 (0.94) | -0.79 (0.88)

21. Secondary Outcome: Change From Baseline in Number of Inhalations Per Day of Salbutamol/Albuterol or Levosalbutamol/Levalbuterol for Symptom Relief at Weeks 48 and 96: Participants From Study DRI12544
Description: The number of salbutamol/albuterol or levosalbutamol/levalbuterol inhalations was recorded daily by the participants in an electronic diary/PEF meter. Mean number of inhalations in last 7 days prior to each visit was calculated and was used in computation of data reported. For this analysis, baseline was defined as parent DRI12544 study baseline.
Time Frame: Baseline of parent study, Week 48, and Week 96 of this extension study
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: inhalations per day
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421
inhalations per day
  Week 48: number analyzed (Participants) | 108 | 406
  Week 48 | -0.00 (3.65) | 0.68 (4.80)
  Week 96: number analyzed (Participants) | 88 | 325
  Week 96 | -0.14 (4.17) | -0.82 (5.18)

22. Secondary Outcome: Change From Baseline in Number of Nocturnal Awakenings at Weeks 48 and 96: Participants From Study DRI12544
Description: The number of nocturnal awakening because of asthma symptoms were recorded every morning by the participants in an electronic diary. Mean number of awakenings in last 7 days prior to each visit was calculated and was used in computation of data reported. For this analysis, baseline was defined as parent DRI12544 study baseline.
Time Frame: Baseline of parent study, Week 48 and Week 96 of this extension study
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: nocturnal awakenings
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421
nocturnal awakenings
  Week 48: number analyzed (Participants) | 110 | 410
  Week 48 | -0.27 (0.54) | -0.43 (0.89)
  Week 96: number analyzed (Participants) | 92 | 344
  Week 96 | -0.29 (0.58) | -0.49 (0.96)

23. Secondary Outcome: Percent Change From Baseline in Oral Corticosteroid (OCS) Dose at Weeks 48, and 96: Participants From Study EFC13691
Description: OCS was allowed as background controller medication for the participants from study EFC13691 only. For this analysis, baseline was defined as parent study EFC13691 baseline.
Time Frame: Baseline of parent study, Weeks 48 and 96 of this extension study
Population: Analysis was performed on exposed population. Here, 'number analyzed' = number of participants with available data for each specified category. Data were planned to be collected and analyzed only for the participants from Study EFC13691 and not for the participants from other studies.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab
Number analyzed (Participants) | 97 | 90
percent change
  Week 48: number analyzed (Participants) | 77 | 57
  Week 48 | 55.32 (42.98) | 80.23 (30.44)
  Week 96: number analyzed (Participants) | 28 | 19
  Week 96 | 71.37 (29.37) | 88.16 (26.83)

24. Secondary Outcome: Percentage of Participants Achieving a Reduction of 50% or Greater (≥ 50% ) in OCS Dose Over Time at Weeks 48 and 96: Participants From Study EFC13691
Description: OCS was allowed as background controller medication for the participants from study EFC13691 only. Percentage of participants who achieved a reduction of ≥ 50% in OCS dose were reported.
Time Frame: Weeks 48 and 96 of this extension study
Population: as for outcome 23
Measure: Number; unit: percentage of participants
Arm/Group | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab
Number analyzed (Participants) | 97 | 90
percentage of participants
  Week 48: number analyzed (Participants) | 77 | 57
  Week 48 | 64.9 | 86.0
  Week 96: number analyzed (Participants) | 28 | 19
  Week 96 | 82.1 | 94.7

25. Secondary Outcome: Percentage of Participants With Background OCS Completely Tapered Off Over Time at Weeks 48 and 96: Participants From Study EFC13691
Description: OCS was allowed as background controller medication for the participants from study EFC13691 only. Number of participants who gradually discontinued or reduced therapeutic dose were reported in this outcome measure.
Time Frame: Weeks 48, and 96 of this extension study
Population: as for outcome 23
Measure: Number; unit: percentage of participants
Arm/Group | Participants From EFC13691: Placebo/Dupilumab | Participants From EFC13691: Dupilumab/Dupilumab
Number analyzed (Participants) | 97 | 90
percentage of participants
  Week 48: number analyzed (Participants) | 77 | 57
  Week 48 | 31.2 | 59.6
  Week 96: number analyzed (Participants) | 28 | 19
  Week 96 | 42.9 | 78.9

26. Secondary Outcome: Change From Baseline in European-Quality of Life-5 Dimension Instrument-3 Levels (EQ-5D-3L) Index Scores at Weeks 48 and 96: Participants From Study DRI12544
Description: EQ-5D-3L: validated and reliable self-report health status questionnaire consisted of EQ-5D descriptive system and visual analogue scale (VAS). EQ-5D descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension measured on 3 levels: no problem, some problems, and severe problems. The 5 dimensional 3-level systems was converted into single index utility score, and the score was 0 - 100, where 100=best health state; and 0=worst health state; where higher scores indicated better outcome. For this analysis, baseline was defined as parent DRI12544 study baseline.
Time Frame: Baseline of parent study, Week 48 and Week 96 of this extension study
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421
score on a scale
  Week 48: number analyzed (Participants) | 100 | 370
  Week 48 | 0.13 (0.20) | 0.14 (0.21)
  Week 96: number analyzed (Participants) | 69 | 294
  Week 96 | 0.12 (0.18) | 0.13 (0.21)

27. Secondary Outcome: Change From Baseline in EQ-5D-3L VAS Scores at Weeks 48 and 96: Participants From Study DRI12544
Description: EQ-5D VAS was used to record a participant's rating for his/her current health-related quality of life state and captured on a vertical VAS (0-100), where 0=worst imaginable health state and 100=best imaginable health state, where higher states indicated better outcomes. For this analysis, baseline was defined as parent DRI12544 study baseline.
Time Frame: Baseline of parent study, Week 48 and Week 96 of this extension study
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants From DRI12544: Placebo/Dupilumab | Participants From DRI12544: Dupilumab/Dupilumab
Number analyzed (Participants) | 111 | 421
score on a scale
  Week 48: number analyzed (Participants) | 100 | 370
  Week 48 | 10.10 (15.40) | 12.88 (18.76)
  Week 96: number analyzed (Participants) | 69 | 294
  Week 96 | 9.90 (18.92) | 13.95 (18.81)

ADVERSE EVENTS:
Time Frame: Reported AE and deaths were TEAEs that developed, worsened, or became serious and deaths that occurred during the TEAE period (time from the first dose of dupilumab in LTS12551 up to the last dose of dupilumab plus 14 weeks) (i.e. up to 108 weeks).
Description: Analysis was performed on safety population.
Groups:
- Participants From DRI12544 Study Placebo/Dupilumab: Participants who completed treatment of placebo (for dupilumab) and post-treatment period in study DRI12544, received a loading dose of dupilumab 600 mg on Day 1 followed by a SC dose of dupilumab 300 mg q2w for 96 weeks in combination with ICS therapy/LABA therapy in this extension study. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Participants From DRI12544 Study Dupilumab/Dupilumab: Participants who completed the treatment of dupilumab and post-treatment period in study DRI12544, received a loading dose of dupilumab 600 mg on Day 1 followed by a SC dose of dupilumab 300 mg q2w for 96 weeks in combination with ICS therapy/LABA therapy in this extension study. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Participants From EFC13579 Study Placebo/Dupilumab: Participants who completed the treatment of placebo (for dupilumab) in study EFC13579 and, who were enrolled before amendment 4 received a SC dose of dupilumab 300 mg q2w for 96 weeks and those who were enrolled after amendment 4 received a SC dose of dupilumab 300 mg q2w for 48 weeks in combination with ICS therapy/LABA therapy in this extension study. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Participants From EFC13579 Study Dupilumab/Dupilumab: Participants who completed the treatment for dupilumab in study EFC13579 and, who were enrolled before amendment 4 received a SC dose of dupilumab 300 mg q2w for 96 weeks and those who were enrolled after amendment 4 received a SC dose of dupilumab 300 mg q2w for 48 weeks in combination with ICS therapy/LABA therapy in this extension study. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Participants From EFC13691 Study Placebo/Dupilumab: Participants who completed the treatment of placebo (for dupilumab) in study EFC13691 and, who were enrolled before amendment 4 received a SC dose of dupilumab 300 mg q2w for 96 weeks and those who were enrolled after amendment 4 received a SC dose of dupilumab 300 mg q2w for 48 weeks in combination with OCS and ICS therapy in this extension study. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Participants From EFC13691 Study Dupilumab/Dupilumab: Participants who completed the treatment of dupilumab in study EFC13691 and, who were enrolled before amendment 4 received a SC dose of dupilumab 300 mg q2w for 96 weeks and those who were enrolled after amendment 4 received a SC dose of dupilumab 300 mg q2w for 48 weeks in combination with OCS and ICS therapy in this extension study. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Participants From PDY14192 Study Placebo/Dupilumab: Participants who completed the treatment of placebo (for dupilumab) in study PDY14192 received a SC dose of dupilumab 300 mg q2w for up to 96 weeks in combination with CS therapy in this extension study. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
- Participants From PDY14192 Study Dupilumab/Dupilumab: Participants who completed the treatment of dupilumab in study PDY14192, received a SC dose of dupilumab 300 mg q2w for up to 96 weeks in combination with ICS therapy in this extension study. Salbutamol/albuterol or Levosalbutamol/levalbuterol was given as reliever medication.
Arm/Group | Participants From DRI12544 Study Placebo/Dupilumab | Participants From DRI12544 Study Dupilumab/Dupilumab | Participants From EFC13579 Study Placebo/Dupilumab | Participants From EFC13579 Study Dupilumab/Dupilumab | Participants From EFC13691 Study Placebo/Dupilumab | Participants From EFC13691 Study Dupilumab/Dupilumab | Participants From PDY14192 Study Placebo/Dupilumab | Participants From PDY14192 Study Dupilumab/Dupilumab
All-Cause Mortality (participants affected / at risk) | 0/111 | 3/421 | 0/517 | 1/1013 | 0/97 | 0/90 | 0/19 | 0/14
Serious Adverse Events (participants affected / at risk) | 14/111 | 42/421 | 48/517 | 106/1013 | 12/97 | 10/90 | 0/19 | 4/14
Other Adverse Events (participants affected / at risk) | 80/111 | 323/421 | 357/517 | 666/1013 | 56/97 | 55/90 | 18/19 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants From DRI12544 Study Placebo/Dupilumab (N=111) | Participants From DRI12544 Study Dupilumab/Dupilumab (N=421) | Participants From EFC13579 Study Placebo/Dupilumab (N=517) | Participants From EFC13579 Study Dupilumab/Dupilumab (N=1013) | Participants From EFC13691 Study Placebo/Dupilumab (N=97) | Participants From EFC13691 Study Dupilumab/Dupilumab (N=90) | Participants From PDY14192 Study Placebo/Dupilumab (N=19) | Participants From PDY14192 Study Dupilumab/Dupilumab (N=14)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Left Ventricular Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina Unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2) | 5 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular Block Complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial Ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odontogenic Cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angle Closure Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serous Retinal Detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Incarcerated Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diaphragmatic Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulum Intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis Erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis Eosinophilic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-Abdominal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large Intestine Polyp (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal Food Impaction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneum Cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adverse Drug Reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic Granulomatosis With Polyangiitis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess Limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary Aspergillosis Allergic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes Simplex Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large Intestine Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mycobacterium Avium Complex Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 4 (4) | 4 (4) | 7 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post Procedural Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chemical Peritonitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Forearm Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incision Site Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional Hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post Procedural Constipation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign Ovarian Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibroadenoma Of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Follicular Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Juvenile Melanoma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large Intestine Benign Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid Artery Disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive Cerebrovascular Disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Idiopathic Intracranial Hypertension (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic Neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parkinson's Disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thalamic Infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed Mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iga Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal Prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 13 (13) | 18 (19) | 0 (0) | 5 (5) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Septum Perforation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis Noninfective (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Status Asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vocal Cord Polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash Vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miscarriage Of Partner (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic Dilatation (Vascular disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants From DRI12544 Study Placebo/Dupilumab (N=111) | Participants From DRI12544 Study Dupilumab/Dupilumab (N=421) | Participants From EFC13579 Study Placebo/Dupilumab (N=517) | Participants From EFC13579 Study Dupilumab/Dupilumab (N=1013) | Participants From EFC13691 Study Placebo/Dupilumab (N=97) | Participants From EFC13691 Study Dupilumab/Dupilumab (N=90) | Participants From PDY14192 Study Placebo/Dupilumab (N=19) | Participants From PDY14192 Study Dupilumab/Dupilumab (N=14)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 0 (0) | 4 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 12 (13) | 9 (11) | 13 (16) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 5 (5) | 6 (6) | 10 (11) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 1 (2) | 6 (6) | 4 (4) | 9 (9) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 16 (20) | 7 (9) | 25 (27) | 4 (4) | 3 (3) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 7 (8) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 13 (14) | 13 (15) | 21 (23) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 6 (36) | 8 (8) | 14 (52) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (4) | 5 (5) | 13 (15) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Fatigue (General disorders) | 1 (1) | 10 (12) | 5 (5) | 8 (15) | 5 (5) | 1 (1) | 0 (0) | 1 (1)
Injection Site Bruising (General disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site Erythema (General disorders) | 26 (102) | 55 (412) | 35 (148) | 50 (295) | 5 (12) | 2 (29) | 8 (21) | 6 (29)
Injection Site Haematoma (General disorders) | 4 (4) | 2 (2) | 4 (4) | 4 (7) | 1 (3) | 0 (0) | 0 (0) | 2 (2)
Injection Site Haemorrhage (General disorders) | 5 (7) | 5 (5) | 5 (5) | 2 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection Site Oedema (General disorders) | 4 (9) | 14 (84) | 14 (32) | 15 (58) | 0 (0) | 2 (8) | 3 (6) | 2 (4)
Injection Site Pain (General disorders) | 9 (18) | 18 (28) | 15 (40) | 14 (51) | 0 (0) | 2 (9) | 1 (3) | 2 (2)
Injection Site Pruritus (General disorders) | 12 (23) | 16 (54) | 15 (36) | 7 (20) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Injection Site Reaction (General disorders) | 0 (0) | 1 (1) | 3 (3) | 5 (10) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection Site Warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (20) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral Swelling (General disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 8 (12) | 0 (0) | 16 (20) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Multiple Allergies (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 15 (30) | 80 (135) | 63 (100) | 117 (181) | 9 (10) | 14 (15) | 0 (0) | 0 (0)
Bronchitis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 5 (5) | 5 (5) | 18 (21) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 6 (6) | 7 (8) | 10 (14) | 26 (31) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Genital Herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 5 (5) | 44 (52) | 30 (39) | 67 (79) | 9 (11) | 7 (10) | 2 (2) | 2 (2)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (2) | 6 (6) | 6 (7) | 17 (18) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 27 (47) | 109 (208) | 99 (149) | 191 (293) | 17 (30) | 16 (22) | 3 (8) | 6 (8)
Oral Candidiasis (Infections and infestations) | 1 (5) | 9 (19) | 6 (9) | 14 (19) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 16 (21) | 37 (57) | 26 (30) | 59 (75) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 0 (0) | 1 (2) | 6 (6) | 7 (7) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Post Procedural Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulpitis Dental (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 3 (3) | 15 (17) | 5 (6) | 18 (25) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 3 (6) | 6 (7) | 11 (15) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 7 (8) | 11 (11) | 6 (7) | 22 (25) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 9 (16) | 33 (56) | 32 (43) | 50 (66) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 18 (30) | 60 (87) | 65 (96) | 130 (213) | 8 (12) | 6 (15) | 2 (4) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 5 (7) | 26 (31) | 17 (20) | 42 (53) | 4 (4) | 3 (3) | 0 (0) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 2 (3) | 11 (15) | 13 (16) | 30 (48) | 1 (4) | 1 (3) | 1 (1) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 6 (9) | 40 (44) | 28 (31) | 45 (48) | 5 (5) | 5 (6) | 2 (2) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 2 (2) | 4 (5) | 3 (3) | 9 (9) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 14 (27) | 12 (13) | 14 (18) | 0 (0) | 2 (3) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 7 (8) | 12 (12) | 33 (38) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Intentional Overdose (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 3 (3) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Lip Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 10 (10) | 7 (7) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Stab Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth Fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Glucose Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
C-Reactive Protein Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epstein-Barr Virus Test Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White Blood Cells Urine Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 23 (29) | 23 (29) | 22 (22) | 7 (7) | 1 (1) | 0 (0) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 30 (33) | 23 (28) | 52 (67) | 5 (5) | 0 (0) | 2 (2) | 3 (4)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6) | 3 (3) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (6) | 7 (9) | 9 (10) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 14 (14) | 7 (7) | 12 (14) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 7 (8) | 16 (16) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (4) | 0 (0) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 12 (13) | 8 (8) | 6 (7) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 13 (14) | 47 (141) | 47 (69) | 74 (145) | 4 (4) | 5 (5) | 4 (9) | 1 (1)
Migraine (Nervous system disorders) | 2 (2) | 3 (3) | 7 (14) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 4 (6) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 7 (7) | 10 (11) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (3) | 6 (7) | 6 (6) | 8 (8) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sleep Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 16 (24) | 10 (12) | 22 (29) | 3 (3) | 3 (4) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 10 (11) | 8 (8) | 12 (23) | 2 (7) | 2 (3) | 2 (2) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 3 (3) | 5 (5) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 13 (13) | 11 (11) | 20 (22) | 2 (2) | 5 (5) | 1 (1) | 1 (1)
Paranasal Sinus Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sputum Increased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (5) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5) | 5 (5) | 9 (11) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyshidrotic Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papulopustular Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pityriasis Alba (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash Generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Solar Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 16 (19) | 19 (20) | 29 (37) | 5 (7) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT02134028/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT02134028/SAP_001.pdf